CLINICAL TRIAL: NCT01321086
Title: Promoting Walking in African Americans With Peripheral Arterial Disease
Brief Title: Motivational Interviewing (MI) for African Americans With Peripheral Arterial Disease (PAD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Tracie Collins, MD, MPH, Preventive Medicine and Public Health Chair, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 7R01HL098909-03 (NIH); 7R01HL098909-03 (NIH)
Record Dates: First submitted 2011-02-16; First posted 2011-03-23 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Peripheral Arterial Disease
Keywords: PAD
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Motivational Interviewing (Active Comparator): Motivational Interviewing (MI) is an effective counseling method in individuals who are less ready to change their behavior. 9 MI sessions will be conducted over the course of the six month intervention.
  Interventions: Behavioral: Motivational Interviewing
- PACE (Active Comparator): Patient-centered Assessment and Counseling for Exercise (PACE) is a protocol that targets known modifiable determinants of behavior change to motivate participants to increase their physical activity (walking).
  Interventions: Behavioral: PACE
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Motivational Interviewing — 9 sessions of MI from baseline to six months
  Arms: Motivational Interviewing
Behavioral: PACE — 9 sessions of PACE delivered from baseline to six months
  Arms: PACE

SUMMARY:
The investigators are conducting a clinical research trial to determine the role of motivational interviewing (MI) on promoting home-based walking therapy to improve walking ability in African Americans with peripheral arterial disease (PAD). African Americans are more than two times as likely as non-Hispanic whites to suffer from PAD. For patients with PAD, there is a significant risk for poor walking ability and limb loss. One major treatment for PAD is walking therapy but the traditional methods for the delivery of this treatment have required frequent visits to a university or hospital-based site. The investigators will address the role of self-managed walking program, to be conducted at or near the home, to improve limb function. In order to motivate the participants to walk, the investigators included two different intervention strategies: MI and patient-centered counseling for exercise (PACE). The investigators hypothesize that participants randomized to the MI arm will have a greater increase in their walking distance, compared to those receiving Patient-Centered Assessment and Counseling for Exercise (PACE) and the control group.

DETAILED DESCRIPTION:
MI is an effective counseling method in individuals who are less ready to change their behavior (i.e., low motivation). Thus, MI is an ideal counseling method to promote home-based walking among AAs with PAD. In our pilot study to promote home-based walking, we used a counseling protocol, Patient-centered Assessment and Counseling for Exercise (PACE)(Sallis et al), which targets known modifiable determinants of behavior change (e.g., social support). Using PACE, we demonstrated an improvement in stair climbing ability and lower limb blood flow (as measured by the ankle-brachial index). Improvements in these lower limb outcomes offer support for the use of PACE counseling in PAD, but PACE does not specifically address low motivation - a critical target for AAs with PAD. In addition, PACE is not culturally sensitive. In our proposed trial, we hypothesize that MI will improve walking distance and reduce walking impairment more than PACE in AAs with PAD.

There is a critical need to improve lower limb outcomes in AAs with PAD. Our long-term goal is to reduce debilitating functional limitations and amputations in AAs with PAD. The overall objective of this application is to determine the most effective counseling strategy to improve home-based walking in AAs with PAD. We have assembled an excellent and diverse research team with the requisite skills and experience needed for this study. Moreover, we have robust pilot data to support the study hypotheses and ensure successful completion of the study.

We will deliver the PACE protocol or MI for 6 months, using both face-to-face visits and telephone contact. Our primary outcome is walking distance (as measured by the widely used and well-validated 6-minute walk test) at the end of active intervention (6 months). Secondary outcomes are walking distance as measured beyond the active phase of intervention (12 months), use of home-based walking (as measured by accelerometry), and lower limb blood flow (as measured by the ankle brachial index - ABI). Our comparison group will receive the same print material as the two interventions as well as contact every three months to update any changes in contact information and to assess their health status. We will randomize 204 participants to one of three arms: Control or Treatment One (Tx1); PACE or Treatment Two (Tx2); or MI, also referred to as Treatment Three (Tx3). In addition, we will determine the efficacy of PACE (Tx2) to increase walking distance in AAs with PAD, compared to Control (Tx1).

Primary Hypothesis:

1. At 6 months, AAs with PAD randomized to MI (Tx3) will have a greater increase in their walking distance, compared to those receiving PACE (Tx2) and the control group (Tx1).

Secondary Hypotheses:

1. AAs with PAD randomized to MI (Tx3) will have a greater increase in their walking distance at 12 months - a follow-up period beyond the six months of active intervention - compared to those receiving PACE (Tx2) and compared to the control group (Tx1).
2. At 6 and 12 months, AAs with PAD randomized to MI (Tx3) will have a greater increase in their home-based walking and their lower limb blood flow, compared to those receiving PACE (Tx2) and to the control group (Tx1).
3. At 6 and 12 months, AAs with PAD randomized to PACE (Tx2) will have a greater increase in their walking distance compared to those randomized to control (Tx1).

Exploratory Aim:

We will explore potential mediators (self-efficacy, social support, intrinsic/extrinsic motivation) and moderators (co-morbidities, leg symptom type, stage of change) of intervention effects on walking distance, home-based walking, and lower limb blood flow among AAs with PAD.

ELIGIBILITY:
Inclusion Criteria:

1. African American (determined by self-report)
2. Lived most of their life in the United States
3. Resting ABI <0.995
4. English Speaking
5. Has a telephone

Exclusion Criteria:

1. Currently walking for exercise at least 5 days per week (i.e., a PACE score ranging from 5-8); the rationale is that a person who is currently walking for at least 5 days per week is already sufficiently active and therefore not a member of the target population for our motivational home-based walking intervention.
2. Prior major amputation (foot or lower leg) or critical leg ischemia (tissue loss, gangrene, or ulcers)
3. Rest pain with ABI <0.4 and non-palpable femoral pulses without prior evaluation by a vascular surgeon, given the need for evaluation for the role of more invasive therapy prior to recommending walking therapy
4. Leg revascularization within 3 months of enrollment or plans for revascularization during the study period; the rationale is that post intervention recovery and potential complications are likely to limit the patient's ability to adhere to the study protocol.
5. Use of supplemental oxygen; the rationale for this is concern for participant safety and potential limited ability to participate in the study secondary to breathing difficulty.
6. Myocardial infarction within the preceding 3 months; the rationale for this is participant safety and the potential risk for complications and/or the need for supervised cardiac rehabilitation following the event.
7. Resting blood pressure > 200/110 mmHg; the rationale for this is participant safety, as blood pressure may further increase during exercise and increase risk for a cerebrovascular event or myocardial infarction.
8. Exercise-induced coronary ischemic symptoms, or exercise-induced ST depression > 2.0 mm; the rationale for this is participant safety and the need for further cardiac evaluation prior to involvement in walking therapy (American College of Cardiology/American Heart Association, 2006).
9. Inability to walk for 2 minutes; the rationale being that people who cannot walk for 2 minutes would not be able to complete the necessary submaximal treadmill test, which is used to screen for coronary ischemic symptoms. We will also exclude anyone who can walk for 20 minutes or more during the submaximal treadmill test. Anyone who can complete the submaximal test would not have significant walking impairment and would not get that much out of the study. Short Physical Performance Battery score of 10 or higher as such persons do not have a clinically significant impairment in mobility; therefore, we will exclude anyone who scores a 10 or higher (out of a maximum of 12 points).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2011-06; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
6 Minute Walk Test | 6 months
  Distance walked in 6 minutes

SECONDARY OUTCOMES:
Short Physical Performance Battery (SPPB) | Baseline
  Assessment of balance and basic physical mobility
Blood work for glucose and lipid levels | Baseline
  glycosylated hemoglobin (HbA1C) and a fasting lipid profile
Adherence to Physical Activity | Baseline
  The participants will be asked to wear accelerometers for seven days at each of the three time points.
Ankle-Brachial Index (ABI) | Baseline
  An assessment that is used to determine the severity of peripheral arterial disease.
Quality of Life | Baseline
  The SF-12 and VascQOL questionnaires will be used to assess QOL.
6 minute walk test | 12 months
  Distance walked in 6 minutes
6 minute walk test | Baseline
  Distance walked in 6 minutes
Short physical performance battery (SPPB) | 6 months
  Assessment of balance and basic physical mobility
Short Physical Performance Battery (SPPB) | 12 months
  Assessment of balance and basic physical mobility
Blood work for glucose and lipid levels | 6 months
  HbA1C and a fasting lipid profile
Blood work for glucose and lipid levels | 12 months
  HbA1C and a fasting lipid profile
Ankle-Brachial Index (ABI) | 12 months
  An assessment that is used to determine the severity of peripheral arterial disease.
Quality of Life | 6 months
  The SF-12 and VascQOL questionnaires will be used to assess QOL.
Quality of life | 12 months
  The SF-12 and VascQOL questionnaires will be used to assess QOL.
Dietary habits for fats and fruits and vegetables | baseline
  Assessment of fats and fruit and vegetable intake
Dietary habits for fats and fruits and vegetables | 6 months
  Assessment of fats and fruit and vegetable intake
Dietary habits for fats and fruits and vegetables | 12 months
  Assessment of fats and fruit and vegetable intake
Adherence to Physical Activity | 6 months
  The participants will be asked to wear accelerometers for seven days at each of the three time points.
Adherence to Physical Activity | 12 months
  The participants will be asked to wear accelerometers for seven days at each of the three time points.

CONTACTS AND LOCATIONS:
Overall Officials: Tracie C Collins, MD, MPH, Principal Investigator — KU School of Medicine-Wichita
Locations (2):
- United States (2):
  - Clinical and Translational Science Unit, Fairway, Kansas
  - KU School of Medicine-Wichita, Wichita, Kansas

REFERENCES:
- [Derived] Collins TC, Lu L, Ahluwalia JS, Nollen NL, Sirard J, Marcotte R, Post S, Zackula R. Efficacy of Community-Based Exercise Therapy Among African American Patients With Peripheral Artery Disease: A Randomized Clinical Trial. JAMA Netw Open. 2019 Feb 1;2(2):e187959. doi: 10.1001/jamanetworkopen.2018.7959. PMID 30768192
- [Derived] Love B, Nwachokor D, Collins T. Recruiting African Americans with peripheral artery disease for a behavioral intervention trial. Vasc Med. 2016 Aug;21(4):345-51. doi: 10.1177/1358863X16628646. Epub 2016 Feb 18. PMID 26893320